CLINICAL TRIAL: NCT00291837
Title: Phase II Open Label Study of CT-2106 as a Single Agent in Patients With Advanced Metastatic Ovarian Cancer Who Have Failed One Prior Platinum and Taxane Based Regimen
Brief Title: CT-2106 for the Second Line Treatment of Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM203
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian; CT-2106
MeSH Terms: conditions — Ovarian Neoplasms | interventions — polyglutamate camptothecin

INTERVENTIONS:
Drug: CT-2106

SUMMARY:
The purpose of this sudy is to determine the response rate of CT-2106 in patients with advanced ovarian cancer who have failed one prior platinum and taxane based regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced ovarian carcinoma, who have failed one prior platinum and taxane containing regimen
* Only one prior chemotherapy containing either cisplatin or carboplatin plus taxanes administered concomitantly
* At least one measurable lesion according to RECIST
* ECOG performance status 0 or 1
* at least 18 years old
* Adequate haematological function
* Adequate renal and hepatic functions
* Normal coagulation parameters

Exclusion Criteria:

* Platinum-sensitive patients (Group 2) who responded (CR or PR) to a 1st line therapy and subsequently progressed or relapsed after a treatment-free interval of > 12 months
* Pregnant or lactating patients
* Prior treatment with camptothecins
* Presence or history of CNS metastasis or carcinomatous leptomeningitis;
* Current active infection per investigator assessment;
* Unresolved bowel obstruction or subobstruction, uncontrolled Crohn's disease or ulcerative colitis;
* Current history of chronic diarrhea >= grade 1 (CTCAE version 3);
* Surgery or radiotherapy ≤ 4 weeks before first study treatment. In case of cytoreductive surgery for the progression of the disease, ≤ 2 weeks before the 1st study treatment are allowed;
* Other uncontrolled, serious illness or medical condition, as determined by the investigator;
* Concomitant (or within 4 weeks before inclusion) administration of any other experimental drug under investigation;
* Concurrent treatment with any other anti-cancer therapy;
* Known HIV positivity or AIDS-related illness;
* Patients who cannot be regularly followed up for psychological, social, familial or geographic reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-11; Primary Completion 2006-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
toxicity
response duration
time to progression
survival

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Calvert, PhD, Principal Investigator — Newcastle General Hospital
Locations (7):
- France (2):
  - Lyon
  - Saint-Brieuc
- Campobasso, Italy
- United Kingdom (4):
  - Birmingham
  - London
  - Newcastle upon Tyne
  - Surrey